CLINICAL TRIAL: NCT04563039
Title: Evaluation of Applaud Medical's Acoustic Enhancer With Laser Lithotripsy System in the Treatment of Urinary Stones
Brief Title: Acoustic Enhancer Research on Laser Lithotripsy (AEROLITH)
Acronym: AEROLITH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avvio Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIP-0001
Record Dates: First submitted 2020-09-15; First posted 2020-09-24 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Urinary Stones
Keywords: Fragmentation of calcium-based urinary stones; Fragmentation of urinary stones
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Intervention Model Description: This study is a double blinded study in which study subjects will not be informed of their treatment allocation through the index procedure. In assessing stone fragmentation using a CT image as defined in the primary endpoint, an independent radiologist will conduct the assessment and will be blinded to the treatment allocation of each subject's CT image.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Ureteroscopic Laser Lithotripsy with Acoustic Enhancer (Experimental): Ureteroscopic Laser Lithotripsy with Acoustic Enhancer
  Interventions: Device: Ureteroscopy Laser Lithotripsy (URS-LL) with Acoustic Enhancer
- Standard Ureteroscopic Laser Lithotripsy (Active Comparator): Standard Ureteroscopic Laser Lithotripsy
  Interventions: Device: Standard Ureteroscopic Laser Lithotripsy

INTERVENTIONS:
Device: Ureteroscopy Laser Lithotripsy (URS-LL) with Acoustic Enhancer — Applaud's Acoustic Enhancer is provided in a lyophilized form. After reconstitution, it is a liquid, containing micron-scale particles that are made of a perfluoroalkane gas core with a lipid shell. The device is intended to be used with cleared/approved pulsed laser systems in fragmenting urinary stones (calculi) in the upper (superior) pole, lower (inferior) pole, and interpolar region of the kidney, pelvis of the kidney, and proximal ureter.
  Arms: Ureteroscopic Laser Lithotripsy with Acoustic Enhancer
Device: Standard Ureteroscopic Laser Lithotripsy — Standard of care Ureteroscopic Laser Lithotripsy
  Arms: Standard Ureteroscopic Laser Lithotripsy

SUMMARY:
A pivotal study to evaluate the safety and effectiveness of Applaud Acoustic Enhancer when used in conjunction with conventional ureteroscopic laser lithotripsy (URS-LL) in the treatment of subjects with urinary stones.

DETAILED DESCRIPTION:
The AEROLITH Clinical Study will evaluate the safety and effectiveness of Applaud Acoustic Enhancer when used in conjunction with conventional ureteroscopic laser lithotripsy (URS-LL) in the treatment of subjects with urinary stones. The clinical study is a prospective, multi-center, two-arm, randomized, double blinded study.

A total of 196 subjects will be enrolled in this study at up to 27 investigational sites located in the U.S.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years to ≤ 75 years
2. Provides written informed consent
3. Patients with at least one urinary stone measuring 6mm or greater (but no more than a cumulative diameter of 20mm) located proximally to the iliac vessels on one side may be treated.
4. Urinary stone(s) should be apparent on a CT scan within 60 days prior to study enrollment. Stone assessment will be conducted using CT imaging following CLIN-0025: AEROLITH IDE Study Screening Guide.
5. Patients with bilateral stones are allowed but only one side may be treated. Only the treated side will be evaluated for safety and effectiveness
6. Patients may enter the study with a stent in place.
7. Patients presenting with absence of a Urinary Tract Infection as confirmed using urinalysis

Exclusion Criteria:

1. Patients with stones exceeding a cumulative diameter of 20mm on the side to be treated. Note: Punctate stones measuring ≤ 2mm do not count in the cumulative diameter limit.
2. Patients with ureteral stones located distal to the iliac vessels on the side to be treated
3. Diagnosis of radiolucent stones (on the side to be treated) on KUB or Scout CT Imaging
4. For patients who have a ureteral stent in place, patient is excluded if stent is calcified or encrusted as verified using standard of care imaging (e.g. KUB X-ray)
5. Patients who have had prior URS-LL within 3 months on the side to be treated at the time of consent.
6. History of cystinuria
7. Urine pH is < 5.5.
8. Patients with known history of recurrent uric acid stones
9. Untreated urinary tract infection (UTI)
10. History of drug-resistant chronic UTI
11. If female, pregnant as confirmed using urine test to be conducted on the day of the procedure.
12. Patient has an American Society of Anesthesiologists (ASA) physical classification level of 4 or greater.
13. Known sensitivity to possible medications used before, during, or after the URS Laser Lithotripsy procedure, including but not limited to the following: sedative agents, general anesthetics, topical anesthetics, and opioid analgesics
14. Stones suspected in calyceal diverticula
15. Horseshoe kidney
16. Congenitally ectopic pelvic kidneys
17. Full staghorn calculi >2cm
18. Patients with elevated serum creatinine > 1.5mg/dl
19. Patients with a solitary kidney
20. Malrotated kidney on the side with urinary stone
21. Duplicated collecting system or duplicated ureters
22. Patients who are currently involved in any investigational drug or device trial or have been enrolled in such trials within 30 days of index procedure
23. Patients who are actively taking antiplatelet and anti-coagulation except low dose aspirin
24. Prostate biopsy within the last 3 months
25. History of radiation therapy of abdomen and pelvis
26. History of urinary tract reconstruction
27. Other factors that the investigator feels would interfere with the participation and completion of the study such as:

    * Inability to provide voluntary consent
    * Inability to understand the clinical investigation or cooperate with investigational procedures
    * Planned relocation or unable to return for required follow-up visits
    * Vulnerable individuals (mentally disabled, physically disabled, prisoner, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Yamut, Study Director — Avvio Medical
Locations (23):
- United States (23):
  - University of Alabama, Birmingham, Alabama
  - Arizona Urology Specialists (Previously Arizona Institute of Urology, PLLC), Tucson, Arizona
  - Arkansas Urology Research Center, Little Rock, Arkansas
  - University of California, Irvine, California
  - University of California, San Diego, California
  - University of California, San Francisco, California
  - University of Florida, Gainesville, Florida
  - University of Miami Health, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Wichita Urology Group, Wichita, Kansas
  - Ocshner LSU Health Shreveport - Regional Urology, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Michigan Institute of Urology, Troy, Michigan
  - Mount Sinai West, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Oregon Health and Sciences University, Portland, Oregon
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Urology San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ureteroscopic Laser Lithotripsy With Acoustic Enhancer | Standard Ureteroscopic Laser Lithotripsy
Started | 103 | 93
Completed | 100 | 90
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ureteroscopic Laser Lithotripsy With Acoustic Enhancer | Standard Ureteroscopic Laser Lithotripsy | Total
Number analyzed (Participants) | 103 | 93 | 196
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 103 | 93 | 196
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 50.8 [21 to 75] | 54.7 [19 to 75] | 52.7 [19 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 46 | 98
  Male | 51 | 47 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 14 | 32
  Not Hispanic or Latino | 85 | 79 | 164
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 103 | 93 | 196
BMI [Mean (Full Range); unit: kg/m^2] | 31.183 [14.2 to 64.58] | 30.785 [19.57 to 61.2] | 30.994 [14.2 to 64.58]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Absence of or Have Residual Fragments Measuring Less </= to 2 mm
Description: Study subjects who present with a complete absence of stones, or have residual fragments measuring less than or equal to 2 mm on the treatment side, as assessed by CT imaging
Time Frame: At 30 days post index procedure
Measure: Number; unit: participants
Arm/Group | Ureteroscopic Laser Lithotripsy With Acoustic Enhancer | Standard Ureteroscopic Laser Lithotripsy
Number analyzed (Participants) | 100 | 90
participants | 41 | 42

ADVERSE EVENTS:
Time Frame: 30 days (+ 14 days)
Description: Follow up period was 30 days (+ 14 days). Only subjects with new or worsening hydronephrosis (from baseline) or ongoing SAEs at day 30 were followed through day 90 (+/- 21 days).
Arm/Group | Ureteroscopic Laser Lithotripsy With Acoustic Enhancer | Standard Ureteroscopic Laser Lithotripsy
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/93
Serious Adverse Events (participants affected / at risk) | 4/103 | 5/93
Other Adverse Events (participants affected / at risk) | 36/103 | 43/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ureteroscopic Laser Lithotripsy With Acoustic Enhancer (N=103) | Standard Ureteroscopic Laser Lithotripsy (N=93)
Infection: Urinary Tract (Renal and urinary disorders) | 4 (6) | 2 (5)
Psychological (Psychiatric disorders) | 0 (0) | 1 (1) — Depression
Pain (Renal and urinary disorders) | 0 (0) | 1 (1) — Flank pain
Pulmonary / respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Bilateral pleural effusions
Infection: Genital urinary (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Orchitis and candida of the scrotum
Steinstrasse (Renal and urinary disorders) | 1 (1) | 0 (0) — Steinstrasse
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ureteroscopic Laser Lithotripsy With Acoustic Enhancer (N=103) | Standard Ureteroscopic Laser Lithotripsy (N=93)
Bleeding / vascular disorders (Vascular disorders) | 0 (0) | 1 (1) — Hematuria with or without clots
Cardiovascular: Other (Cardiac disorders) | 0 (0) | 1 (1) — Acute hypertensive episode
Burns (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Altered bowel patters (Gastrointestinal disorders) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Worsening irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection: Fever (Infections and infestations) | 0 (0) | 1 (1)
Vaginal Yeast Infection (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Infection in the genitourinary system (Infections and infestations) | 4 (4) | 3 (5)
Damage to ureter (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) — Including swelling, scarring, damaged urothelium (ipsilateral)
Ureteral mucosal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
COVID-19 related (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Burning (Renal and urinary disorders) | 1 (1) | 0 (0)
Back pain (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Clot retention (General disorders) | 0 (0) | 1 (1)
Perinephric hematoma (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Pain: Abdominal colic (General disorders) | 1 (1) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain: Discomfort (General disorders) | 1 (1) | 0 (0)
Pain: Dysuria (Renal and urinary disorders) | 3 (3) | 5 (5)
Pain: Flank pain, bilateral (General disorders) | 1 (1) | 0 (0)
Pain: flank pain, ipsilateral (General disorders) | 7 (8) | 6 (7)
Pain: Ipsilateral ureteral pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Pain: stent pain (Renal and urinary disorders) | 2 (2) | 0 (0)
Pain: PACU Right abdominal pain (General disorders) | 0 (0) | 1 (1)
Pain: Other (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Pelvic pain due to malpositioned IUD, identified pre-intervention
Pain: Post-op bladder / pelvic pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Pain: Post-op penile pain (General disorders) | 0 (0) | 1 (1)
Pain: flank pain unspecified laterality (General disorders) | 1 (1) | 0 (0)
Pain: surgical pain (General disorders) | 1 (1) | 1 (1)
Pain: Ureteral meatus (Renal and urinary disorders) | 0 (0) | 1 (1)
Pain involved with stent placement / removal and possible dislodging (General disorders) | 2 (2) | 3 (3)
Pain: renal colic (General disorders) | 1 (1) | 2 (2)
Pain: Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Altered creatinine levels (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 3 (3)
Hydroureter (Renal and urinary disorders) | 0 (0) | 1 (1) — Left-side, moderate
Worsening urinary urge incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder spasms (Renal and urinary disorders) | 0 (0) | 2 (2)
Meateal stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic pressure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT04563039/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT04563039/SAP_001.pdf